CLINICAL TRIAL: NCT03617458
Title: Interventions Against Insulin Resistance in Pulmonary Arterial Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Mayo Clinic (Other); The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Anna Hemnes, Associate Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 180198
Record Dates: First submitted 2018-05-02; First posted 2018-08-06 (Actual); Results first posted 2024-10-16 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Artery Hypertension
Keywords: PAH
MeSH Terms: conditions — Familial Primary Pulmonary Hypertension | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: This is a phase II, 2x2 factorial randomized, blinded trial testing metformin versus placebo and a mHealth intervention (mHealth) versus usual care of 12 weeks.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigators propose a phase II, 2x2 factorial randomized, blinded trial testing metformin versus placebo and a mobile health intervention (mHealth) versus usual care of 12 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Metformin + mHealth Intervention (Active Comparator): Patients will receive active ingredient medicine with mHealth texting platform, which are messages designed to facilitate self-awareness, reinforce step targets, and link physical activity with a reward or memorable cue.
  Subjects will receive metformin 500mg. Patients will titrate the medication as follows: 500mg po daily x 5 days, 500mg po twice a day (BID) x 5 days, 500mg by mouth (po) three times a day (TID) x 5 days,1000mg po BID x 69 days (12 weeks total).
  Interventions: Drug: Metformin; Device: mHealth Intervention
- Placebo + Usual Care (Placebo Comparator): Patient will receive non active medicine and routine medical care.
  Interventions: Drug: Placebo; Device: Usual Care
- Metformin + Usual Care (Active Comparator): Patient will receive active ingredient medicine with routine medical care.
  Subjects will receive metformin 500mg. Patients will titrate the medication as follows: 500mg po daily x 5 days, 500mg po BID x 5 days, 500mg po TID x 5 days,1000mg po BID x 69 days (12 weeks total).
  Interventions: Drug: Metformin; Device: Usual Care
- Placebo + mHealth Intervention (Placebo Comparator): Patient will receive non active medicine and the mHealth texting platform, which are messages designed to facilitate self-awareness, reinforce step targets, and link physical activity with a reward or memorable cue.
  Interventions: Drug: Placebo; Device: mHealth Intervention

INTERVENTIONS:
Drug: Metformin — Metformin is a drug has been on the market for several decades and is considered first line therapy for diabetes mellitus type 2.
  Arms: Metformin + Usual Care; Metformin + mHealth Intervention
Drug: Placebo — A treatment with no active ingredients or therapeutic effect.
  Arms: Placebo + Usual Care; Placebo + mHealth Intervention
Device: mHealth Intervention — Our Health Insurance Portability and Accountability Act (HIPAA) compliant texting platform is linked to the Fitbit Application Program Interface. Real time activity data will be transmitted from the subject's smartphone to our mHealth platform via cellular network.Subjects assigned to the texting arm will receive 3 texts/day in sync with their preferred morning, lunch, and evening leisure schedule, which is defined at enrollment. These texts will use personal, disease-specific, and provider information to deliver 2 types of messages customized to the current step count and sent in equal proportion. Messages are designed to facilitate self-awareness, reinforce step targets, and link physical activity with a reward or memorable cue.
  Arms: Metformin + mHealth Intervention; Placebo + mHealth Intervention
Device: Usual Care — Our HIPAA data will be transmitted from the subject's smartphone to our mHealth platform via cellular network.
  Arms: Metformin + Usual Care; Placebo + Usual Care

SUMMARY:
The primary objective of this study is to determine the impact of two interventions against insulin resistance on the composite endpoint of 10% improvement in baseline six minute walk distance or improvement in World Health Organization (WHO) functional class in humans with pulmonary artery hypertension (PAH).

DETAILED DESCRIPTION:
The investigators propose to test the hypothesis that interventions to improve insulin resistance will improve exercise capacity and World Health Organization (WHO) functional class in PAH. The investigators propose three specific aims to test this 1) A prospective 2x2 factorial design 12-week clinical trial of metformin or placebo and activity intervention or usual care to assess effect on six minute walk and WHO functional class, 2) Assessment of the interventions in Aim 1 in a subset of patients on right ventricle (RV) and peripheral muscle function and lipid content and markers of pulmonary vascular disease to define how these interventions may work in PAH and 3) Identify and prospectively test peripheral blood markers of metformin response in PAH. The broad goals of this work are to demonstrate the efficacy and mechanisms of interventions against insulin resistance in PAH and to identify which patients are most likely to benefit from these interventions, moving to precision medicine in PAH.

The investigators are planning a factorial design trial. Patients will be randomized twice. The first is metformin or placebo and is quadruple randomized. The second is mobile health (mHealth) intervention via texts or standard of care and is not blinded to the patients, but is to the investigator and thus is triple randomized.

ELIGIBILITY:
Inclusion Criteria:• Adults aged 18 or older.

* Diagnosed with idiopathic, heritable, or drug- or toxin-associated pulmonary arterial hypertension (PAH) according to World Health Organization consensus recommendations.
* Stable PAH-specific medication regimen for three months prior to enrollment. Subjects with only a single diuretic adjustment in the prior three months will be included. Adjustments in IV prostacyclin for side effect management are allowed.
* Subjects must own a Bluetooth capable modern smartphone capable of receiving and sending text messages and an active data plan.
* WHO Functional Class I-III
* Ambulatory

Exclusion Criteria:

* Prohibited from normal activity due to wheelchair bound status, bed bound status, reliance on a cane/walker, activity-limiting angina, activity-limiting osteoarthritis, or other condition that limits activity
* Pregnancy
* Diagnosis of PAH etiology other than idiopathic, heritable, or associated with drugs or toxins
* FEV1> or = 65% predicted AND normal chest imaging
* WHO Functional class IV heart failure
* Requirement of > 1 diuretic adjustment in the prior 30 days
* Preferred form of activity is not measured by an activity tracker (swimming, ice skating, stair master, or activities on wheels such as bicycling or rollerblading)
* Type I diabetes mellitus
* Prior diagnosis of cirrhosis
* Untreated hypo- or hyper-thyroidism
* estimated glomerular filtration rate (eGFR) by modification of diet in renal disease (MDRD) <60 milliliters per minute (mL/min)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2018-08-23 (Actual); Primary Completion 2023-09-09 (Actual); Study Completion 2025-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna R Hemnes, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] D'Alonzo GE, Barst RJ, Ayres SM, Bergofsky EH, Brundage BH, Detre KM, Fishman AP, Goldring RM, Groves BM, Kernis JT, et al. Survival in patients with primary pulmonary hypertension. Results from a national prospective registry. Ann Intern Med. 1991 Sep 1;115(5):343-9. doi: 10.7326/0003-4819-115-5-343. PMID 1863023
- [Background] Benza RL, Miller DP, Barst RJ, Badesch DB, Frost AE, McGoon MD. An evaluation of long-term survival from time of diagnosis in pulmonary arterial hypertension from the REVEAL Registry. Chest. 2012 Aug;142(2):448-456. doi: 10.1378/chest.11-1460. PMID 22281797
- [Background] Mathai SC, Puhan MA, Lam D, Wise RA. The minimal important difference in the 6-minute walk test for patients with pulmonary arterial hypertension. Am J Respir Crit Care Med. 2012 Sep 1;186(5):428-33. doi: 10.1164/rccm.201203-0480OC. Epub 2012 Jun 21. PMID 22723290

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occured between 8/23/2018-8/22/2023. Recruitment occurred in clinics at each of the participating sites.
Pre-assignment Details: There was a participant run-in for the fitbit portion of the study. Run-in was a 2-week period.
Groups:
- Metformin + mHealth Intervention: Patients will receive active ingredient medicine with mHealth texting platform, which are messages designed to facilitate self-awareness, reinforce step targets, and link physical activity with a reward or memorable cue.
  Subjects will receive metformin 500mg. Patients will titrate the medication as follows: 500mg po daily x 5 days, 500mg po twice a day (BID) x 5 days, 500mg by mouth (po) three times a day (TID) x 5 days,1000mg po BID x 69 days (12 weeks total).
  Metformin: Metformin is a drug has been on the market for several decades and is considered first line therapy for diabetes mellitus type 2.
  mHealth Intervention: Our Health Insurance Portability and Accountability Act (HIPAA) compliant texting platform is linked to the Fitbit Application Program Interface. Real time activity data will be transmitted from the subject's smartphone to our mHealth platform via cellular network.Subjects assigned to the texting arm will receive 3 texts/day in sync with their preferred morning, lunch, and evening leisure schedule, which is defined at enrollment. These texts will use personal, disease-specific, and provider information to deliver 2 types of messages customized to the current step count and sent in equal proportion. Messages are designed to facilitate self-awareness, reinforce step targets, and link physical activity with a reward or memorable cue.
- Metformin + Usual Care: Patient will receive active ingredient medicine with routine medical care.
  Subjects will receive metformin 500mg. Patients will titrate the medication as follows: 500mg po daily x 5 days, 500mg po BID x 5 days, 500mg po TID x 5 days,1000mg po BID x 69 days (12 weeks total).
  Metformin: Metformin is a drug has been on the market for several decades and is considered first line therapy for diabetes mellitus type 2.
  Usual Care: Our HIPAA data will be transmitted from the subject's smartphone to our mHealth platform via cellular network.
Period: Overall Study
Arm/Group | Metformin + mHealth Intervention | Placebo + Usual Care | Metformin + Usual Care | Placebo + mHealth Intervention
Started | 18 | 17 | 19 | 19
Completed | 15 | 14 | 18 | 19
Not Completed | 3 | 3 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin + mHealth Intervention | Placebo + Usual Care | Metformin + Usual Care | Placebo + mHealth Intervention | Total
Number analyzed (Participants) | 18 | 17 | 19 | 19 | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.4 (17.4) | 46.6 (10.7) | 48.8 (13.7) | 47 (12.2) | 47.5 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 15 | 16 | 53
  Male | 6 | 7 | 4 | 3 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 0 | 2
  Not Hispanic or Latino | 18 | 16 | 18 | 19 | 71
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 0 | 2
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 1 | 1 | 0 | 6
  White | 14 | 15 | 15 | 19 | 63
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 18 | 17 | 19 | 19 | 73

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Six Minute Walk Distance (Meters)
Description: The change in meters walked for the six-minute walk distance from baseline to week 12
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Metformin + mHealth Intervention | Placebo + Usual Care | Metformin + Usual Care | Placebo + mHealth Intervention
Number analyzed (Participants) | 14 | 12 | 16 | 18
meters
  Baseline | 414.5 (87.9) | 461.7 (135.6) | 448.9 (85.9) | 483.0 (85.6)
  12-Week | 457.2 (110.2) | 474.9 (123.6) | 454.8 (112.3) | 485.6 (72.3)

2. Primary Outcome: Change From Baseline to Week 12 in World Health Organization Functional Class (WHO FC)
Description: Change from baseline in WHO functional class at week 12. The World Health Organization (WHO) functional class system was created to define the severity of an individual's symptoms and how they impact on day-to-day activities. The columns represent the randomization assignment and the rows represent if a change in WHO functional class occurred by the participant from baseline to week 12.
Time Frame: baseline and 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin + mHealth Intervention | Placebo + Usual Care | Metformin + Usual Care | Placebo + mHealth Intervention
Number analyzed (Participants) | 16 | 14 | 17 | 18
Participants
  Did not improve Functional Class | 15 | 12 | 14 | 13
  Improved Functional Class by at least 1 | 1 | 2 | 3 | 5

3. Secondary Outcome: Change From Baseline to Week 12 in Body Weight (Kilograms)
Description: Change in body weight as measured by assessing weight in kilograms at baseline and at week 12.
Time Frame: baseline and end of 12 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Change From Baseline to Week 12 in Body Mass Index (BMI)
Description: Change from baseline BMI at week 12. BMI is defined as a measure of body fat based on height and weight that applies to adult men and women.
Time Frame: baseline and end of 12 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Change From Baseline to Week 12 in Absolute Six-Minute Walk Distance (Meters)
Description: Change from baseline six-minute walk test distance (meters) at week 12.
Time Frame: baseline and end of 12 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Change From Baseline to Week 12 in Borg Dyspnea Score
Description: Change from baseline Borg dyspnea score at week 12.
  The Borg dyspnea score is a measure of the physical activity intensity level based on the subject's perceived exertion. Subjects will rate at resting and peak exercise. Targets exercise capacity.
Time Frame: baseline and end of 12 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Change From Baseline to Week 12 in Emphasis-10 Quality of Life Survey Score
Description: Change from baseline Emphasis-10 quality of life survey score at week 12. Survey completed at baseline and 12 weeks.
  The emPHasis-10 is a short and easy questionnaire that consists of 10 items which address breathlessness, fatigue, control and confidence. Each item is scored on a semantic differential six-point scale (0-5), with contrasting adjectives at each end. A total emPHasis-10 score is derived using simple aggregation of the 10 items. emPHasis-10 scores range from 0 to 50, higher scores indicate worse quality of life.
Time Frame: baseline and end of 12 weeks
Reporting Status: Not Posted

8. Secondary Outcome: Change From Baseline to Week 12 in Daily Step Count, as Measured by the Mean Daily Step Count
Description: Change from the baseline mean daily step count at week 12. Data obtained by the mHealth device.
Time Frame: baseline and end of 12 weeks
Reporting Status: Not Posted

9. Secondary Outcome: Change From Baseline to Week 12 in Daily Step Count Goal Attainment, as Measured by the Percentage (%) of Subjects Who Meet Their Daily Step Count Goal
Description: Assess the frequency (% of days) that the daily step target was achieved over time. Data obtained by the mHealth device.
Time Frame: baseline and end of 12 weeks
Reporting Status: Not Posted

10. Secondary Outcome: Change From Baseline to Week 12 in Daily Aerobic Time (Minutes)
Description: Change from baseline daily aerobic time at week 12. Aerobic time is defined as total time in minutes spent walking continuously for > 10 minutes without breaking for > 1 minute.
Time Frame: baseline and end of 12 weeks
Reporting Status: Not Posted

11. Secondary Outcome: Change From Baseline to Week 12 in Total Daily Activity Assessed in Step Counts Per Minute
Description: This variable will be assessed by FitBit and is expressed in step counts per minute. Mean value from the last week in the study will be evaluated and mean change from baseline will be calculated.
Time Frame: baseline and end of 12 weeks
Reporting Status: Not Posted

12. Secondary Outcome: Change From Baseline to Week 12 in Resting Heart Rate (Beats Per Minute)
Description: Monitored regularly using activity tracking device (per second when active, per 5 seconds when inactive). Subject's resting and peak exercise heart rate will also be recorded at baseline and week 12. Targets exercise capacity. Heart rate is expressed as beats per minute.
Time Frame: baseline and end of 12 weeks
Reporting Status: Not Posted

13. Secondary Outcome: Change From Baseline to Week 12 in Homeostatic Model Assessment (HOMA)-Insulin Resistance (IR)
Description: Change from baseline insulin resistance at week 12. Insulin resistance will be quantified using the homeostatic model assessment of insulin resistance (HOMA-IR), which estimates insulin resistance through fasting plasma insulin and glucose ratios. Targets mechanism of improved exercise capacity.
Time Frame: baseline and end of 12 weeks
Reporting Status: Not Posted

14. Secondary Outcome: Number of Participants With Abnormal Laboratory Values of Plasma Estradiol Metabolites
Description: As measured by plasma estradiol in pg/ml, DHEA in mcg/ml, total testosterone in ng/dl, bioavailable testosterone in ng/dl, progesterone in ng/ml, and sex hormone binding globulin (SHBG) in nmol/L at baseline and week 12. These laboratory values will be aggregated to assess the number of participants with abnormal laboratory values.
Time Frame: baseline and end of 12 weeks
Reporting Status: Not Posted

15. Secondary Outcome: Number of Participants With Abnormal Laboratory Values of Urine Estradiol Metabolites
Description: As measured by the laboratory values Estrone (E1), Estradiol (E2), 2-OHE1, 2-OHE2, 2-MeOE1, 2-MeOE2, 4-OHE1, 4-MeOE1, 4-MeOE2, 16a-OHE1, 17-epiE3, Estriol (E3), 16-ketoE2, 16-epiE3 with pM per mg of urine creatinine. These laboratory values will be assessed at baseline and week 12 and then aggregated to assess the number of participants with abnormal laboratory values.
Time Frame: baseline and end of 12 weeks
Reporting Status: Not Posted

16. Secondary Outcome: Number of Participants With Abnormal Laboratory Values of Plasma Lipid Profile
Description: As measured by total cholesterol, triglycerides, high-density lipoprotein cholesterol, low-density lipoprotein cholesterol, and non - high-density lipoprotein cholesterol with mg/dl as the units of measure at baseline and week 12. These laboratory values will be aggregated to assess number of participants with abnormal laboratory values.
Time Frame: baseline and end of 12 weeks
Reporting Status: Not Posted

17. Secondary Outcome: Number of Participants With Abnormal Laboratory Values of Plasma Free Fatty Acid Profiles
Description: As measured by plasma free fatty acid profiles at baseline and week 12. Free fatty acids will be measured in mmol/L. This laboratory value will be assessed by the number of patients with abnormal laboratory values.
Time Frame: baseline and end of 12 weeks
Reporting Status: Not Posted

18. Secondary Outcome: Number of Participants With Abnormal Laboratory Values of Plasma Acylcarnitine Profiles
Description: As measured by plasma acylcarnitine profiles at baseline and week 12. We will be measuring the laboratory values of C2, C3, C3-dicarboxylic, C4, C4- hydroxyl, C4-dicarboxylic, C5, C5:1, C5 - hydroxy, C5-dicarboxylic, C6, C8, C10, C10:1, C10:2, C12, C14, C14:1, C14:2, C14-hydroxy, C16, C16:1, C161:-hydroxy, C16-hydroxy, C18, C18:1, C18:2, C18-hydroxy, C18:1-hydroxy, C18:2-hydroxy in the unit of measure nmol/L. These laboratory values will be aggregated to assess the number of participants with abnormal laboratory values.
Time Frame: baseline and end of 12 weeks
Reporting Status: Not Posted

19. Secondary Outcome: Change From Baseline to Week 12 in Plasma Brain Natriuretic Peptide (BNP) Laboratory Value Measured in pg/ml
Description: Change from baseline B-type natriuretic peptide (BNP) level at week 12. BNP is a marker of myocardial stress which decreases with exercise training and measured in pg/ml. Targets mechanism of improved exercise capacity.
Time Frame: baseline and end of 12 weeks
Reporting Status: Not Posted

20. Secondary Outcome: Change From Baseline to Week 12 in Quadriceps Skeletal Muscle Triglyceride Content, as Measured by % Triglycerides
Description: Change from baseline quadriceps Skeletal Muscle Triglyceride Content at week 12 as measured by % triglycerides.
Time Frame: baseline and end of 12 weeks
Reporting Status: Not Posted

21. Secondary Outcome: Change From Baseline to Week 12 in Quadriceps Skeletal Muscle Fatigue, as Measured by Total Time to Muscle Fatigue During the Muscle Strength and Function Test
Description: Change from baseline quadriceps Skeletal Muscle Fatigue at week 12 as measured by total time to muscle fatigue during the muscle strength and function test.
Time Frame: baseline and end of 12 weeks
Reporting Status: Not Posted

22. Secondary Outcome: Change From Baseline to Week 12 in Quadriceps Skeletal Muscle Strength During the Muscle Strength and Function Test, as Measured by Maximum Contraction Strength
Description: Change from baseline quadriceps Skeletal Muscle Strength during the Muscle Strength and Function Test at week 12 as measured by maximum contraction strength.
Time Frame: baseline and end of 12 weeks
Reporting Status: Not Posted

23. Secondary Outcome: Change From Baseline to Week 12 in Quadriceps Skeletal Muscle Contractile Tissue Cross-sectional
Description: Change from baseline in quadriceps skeletal muscle contractile tissue cross-sectional at week 12 as measured by the relative change in the maximum cross-sectional area of muscle tissue of the quadriceps muscle group, measured in the axial anatomical plane.
Time Frame: baseline and end of 12 weeks
Reporting Status: Not Posted

24. Secondary Outcome: Change From Baseline to Week 12 in RV Myocardial Muscle Triglyceride Content, as Measured by % Triglycerides
Description: Change from baseline in right ventricle Myocardial Muscle Triglyceride Content results at week 12 as measured by % triglycerides.
Time Frame: baseline and end of 12 weeks
Reporting Status: Not Posted

25. Secondary Outcome: Change From Baseline to Week 12 in Tricuspid Annular Plane Systolic Excursion (TAPSE), Expressed in mm.
Description: Change from baseline in Tricuspid Annular Plane systolic Excursion (TAPSE) expressed in mm on echocardiogram results at week 12.
Time Frame: baseline and end of 12 weeks
Reporting Status: Not Posted

26. Secondary Outcome: Change From Baseline in Right Ventricle (RV) and Left Ventricle (LV) Ejection Fraction Values as Assessed by Echocardiogram Results, Expressed in Percentage (%).
Description: Change from baseline in RV and Left Ventricle (LV) Ejection Fraction values on echocardiogram results at week 12 and expressed in percentage (%).
Time Frame: baseline and end of 12 weeks
Reporting Status: Not Posted

27. Secondary Outcome: Change From Baseline in Right Ventricle (RV) Fractional Area, as Assessed by Echocardiogram Results, Expressed in Percentage (%).
Description: Change from baseline in right ventricle Fractional Area on echocardiogram results at week 12 and expressed in percentage (%).
Time Frame: baseline and end of 12 weeks
Reporting Status: Not Posted

28. Secondary Outcome: Change From Baseline in Tricuspid Annular Velocity (S'), as Assessed by Echocardiogram Results, Expressed in cm/Sec
Description: Change from baseline in Tricuspid Annular Velocity (S') on echocardiogram results at week 12 and expressed in cm/sec.
Time Frame: baseline and end of 12 weeks
Reporting Status: Not Posted

29. Secondary Outcome: Change From Baseline in Tricuspid Regurgitant (TR) Velocity, as Assessed by Echocardiogram Results, Expressed in m/Sec.
Description: Change from baseline in Tricuspid Regurgitant (TR) Velocity on echocardiogram results at week 12 and expressed in m/sec.
Time Frame: baseline and end of 12 weeks
Reporting Status: Not Posted

30. Secondary Outcome: Change From Baseline in Estimated Right Ventricle (RV) and Right Atrial (RA) Pressure, as Assessed by Echocardiogram Results, Expressed in mmHg
Description: Change from baseline in the estimated right ventricle and right atrial pressure on echocardiogram results at week 12 and expressed in mmHg.
Time Frame: baseline and end of 12 weeks
Reporting Status: Not Posted

31. Secondary Outcome: Change From Baseline in Right Ventricle (RV) and Left Ventricle (LV) Diastolic Function as Assessed by Doppler Inflow Patterns on Echocardiogram.
Description: Change from baseline in right and left ventricular diastolic function as assessed by Doppler inflow patterns on echocardiogram results at week 12
Time Frame: baseline and end of 12 weeks
Reporting Status: Not Posted

32. Secondary Outcome: Change From Baseline in Right Ventricle (RV) Free Wall Longitudinal Strain, as Assessed by Echocardiogram Results, and Expressed as Percent (%) Change in Myocardial Deformation.
Description: Change from baseline in right ventricle free wall longitudinal strain on echocardiogram results at week 12 and expressed as percent (%) change in myocardial deformation.
Time Frame: baseline and end of 12 weeks
Reporting Status: Not Posted

33. Secondary Outcome: Number of Participants With a Change in Screening Clinical Characteristics
Description: To compare and define the screening clinical characteristics of responders and non-responders to mHealth intervention or no intervention and/or metformin at week 12. We will be taking into account all patient screening data including demographic information, medical history, current medication regimen, physical exam, 6MWT, echocardiogram, MRS, skeletal muscle function test, emphasis-10 survey, WHO functional class, and laboratory values. These results will be aggregated and the results compared to the same characteristics at the end of week 12.
  We will be assessing the number of participants with a change in screening clinical characteristics.
Time Frame: baseline and end of 12 weeks
Reporting Status: Not Posted

34. Secondary Outcome: Number of Patients With Treatment - Emergent Adverse Events (Safety and Tolerability of mHealth Intervention and Drug Treatment in PAH Subjects)
Description: Number of treatment-related adverse events as assessed by telephone calls at baseline, week one, week three, week nine, week twelve, and week seventeen.
Time Frame: baseline and end of 12 weeks
Reporting Status: Not Posted

35. Secondary Outcome: Patient Satisfaction of Treatment Interventions, as Measured by Change in Emphasis-10 Survey Score
Description: We will be assessing patient satisfaction of treatment interventions by looking at the number of participants with an increase or decrease in overall score on the emphasis-10 questionnaire from screening and at the end of 12 weeks.
  The emPHasis-10 is a short and easy questionnaire that consists of 10 items which address breathlessness, fatigue, control and confidence. Each item is scored on a semantic differential six-point scale (0-5), with contrasting adjectives at each end. A total emPHasis-10 score is derived using simple aggregation of the 10 items. EmPHasis-10 scores range from 0 to 50, higher scores indicate worse quality of life.
Time Frame: baseline and end of 12 weeks
Reporting Status: Not Posted

36. Secondary Outcome: Dropout Rate Incidence
Description: To assess the effect of a mHealth intervention or no intervention and/or metformin or placebo on dropout rates over 12 weeks.
Time Frame: baseline and end of 12 weeks
Reporting Status: Not Posted

37. Secondary Outcome: Number of Patients With a PAH-related Hospitalization Incidence
Description: To assess the effect of a mHealth intervention or no intervention and/or metformin or placebo on PAH-related hospitalization incidences over 12 weeks. Number of patients will be assessed.
Time Frame: baseline and end of 12 weeks
Reporting Status: Not Posted

38. Secondary Outcome: Change From Baseline to Week 12 in Patient Medication Regimen, as Measured by Percentage (%) of Subjects With a Change in Medication Regimen
Description: Change from baseline in patient medication regimen at week 12 as measured by percentage (%) of subjects with a change in medication regimen.
Time Frame: baseline and end of 12 weeks
Reporting Status: Not Posted

39. Secondary Outcome: Incidence of Death
Description: To assess the effect of a mHealth intervention or no intervention and/or metformin or placebo on incidence of death over 12 weeks.
Time Frame: baseline to/and 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected over study duration-baseline to 12-weeks.
Arm/Group | Metformin + mHealth Intervention | Placebo + Usual Care | Metformin + Usual Care | Placebo + mHealth Intervention
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/17 | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 5/18 | 3/17 | 1/19 | 1/19
Other Adverse Events (participants affected / at risk) | 9/18 | 7/17 | 14/19 | 9/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin + mHealth Intervention (N=18) | Placebo + Usual Care (N=17) | Metformin + Usual Care (N=19) | Placebo + mHealth Intervention (N=19)
Intravenous Medication Line Malfunction/Infection (Product Issues) | 4 (5) | 0 (0) | 0 (0) | 0 (0) — Any issue with the Hickman Catheter that caused hospitalization was considered serious but non-related.
Biliary Colic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Deemed not study related.
Supraventriculartachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) — Resulted in hospitalizations but deemed not relatable.
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Deemed Non-study Related
Infections requiring Hospitalization (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — Included two events,one with pneumonia and one with an upper respiratory infection. Both deemed not-relatable.
Gastrointestinal Bleed (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Bleed was deemed non-study related.
Clinical Worsening (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Related to routine Catheter procedure. Deemed non-study relatable.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin + mHealth Intervention (N=18) | Placebo + Usual Care (N=17) | Metformin + Usual Care (N=19) | Placebo + mHealth Intervention (N=19)
Gastrointestinal Issues (Gastrointestinal disorders) | 8 (12) | 3 (6) | 10 (14) | 3 (3) — Including issues like bloating, nausea, diarrhea, or discomfort. Deemed not to be serious events
Intravenous Medication Line Malfunction/Infection (Product Issues) | 0 (0) | 2 (2) | 1 (1) | 1 (1) — Deemed not serious or relatable.
Common Pulmonary Hypertension Symptoms (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (3) | 5 (9) — Complications are expected in patient population considering pulmonary hypertension diagnosis. Unrelated to study and expected.
General Infection (General disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) — This included not relatable or serious adverse conditions such as cellulitis or general sore throat.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-12): https://cdn.clinicaltrials.gov/large-docs/58/NCT03617458/Prot_SAP_000.pdf